CLINICAL TRIAL: NCT01500668
Title: Botulinum Toxin for Treatment of Catocholamine Induced Finger Necrosis - a Double Blind Randomized Control Prospective Study.
Brief Title: Botulinum Toxin A for Treatment of Catocholamine Induced Finger Necrosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Amir Herman, Principal Investigator, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHEBA-11-9023-AH-CTIL; 9023-11-SMC (Other Grant/Funding Number: Sheba medical center)
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Catocholamine Induced Finger Necrosis
Keywords: Botox; catocholamine; shock; vasomotor; Vasopressin; botulinum toxin
MeSH Terms: conditions — Shock; Diabetes Insipidus | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator): Injection of 200 units of Botulinum Toxin A (BOTOX) to a treated limb. Each limb will be divided to two levels - arterial arch and digital arteries (near MCP/MTP) levels. In each level 100 units of Botox will be injected in 6 injection points in the proximity of the arteries.
  Interventions: Drug: Botox
- Control (Placebo Comparator): Injection of 0.5cc of normal saline (0.9% NaCl) to each injection site as in the Active drug arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botox — Injection of 200 units of Botulinum Toxin A (BOTOX) to a treated limb. Each limb will be divided to two levels - arterial arch and digital arteries (near MCP/MTP) levels. In each level 100 units of Botox will be injected in 6 injection points in the proximity of the arteries.
  Arms: Treatment
Drug: Placebo — Injection of 0.5cc of normal saline (0.9% NaCl) to each injection site as in the Active drug arm.
  Arms: Control

SUMMARY:
Patients in the intensive care unit (ICU) often require blood pressure support of vasoactive drugs such as amines. Finger necrosis (so called "blue toe syndrome") is a well documented phenomena with incidence reaching as high as 60% in patients receiving vasopressin. Botulinum toxin is a known muscle relaxant used for a variety of medical application. Recently, several reports have demonstrated its effect in vasospastic disorders. It has also been in mice that when administered locally it has a local vasodilatory effect. The goal of this experiment is to compare the effect of Botulinum Toxin administered locally on amine induced finger necrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with vasoactive drugs (amines) and have finger/toe necrosis

Exclusion Criteria:

* Sensitivity to drug (Botox) ingredients.
* Active local limb infection
* ICU admission due to botulism
* Chronic muscular weakness disease, e.g., Myasthenia gravis, ALS
* Age lower than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
index of Toe and Finger Ischemia (iTFI) | three months after drug administration
  Score including:
  O2 peripheral saturation monitoring Bleeding Capillary refilling Limb temperature Limb discoloration

SECONDARY OUTCOMES:
Amputation | Three months after drug administration
  Amputations performed - fingers, toe and limb - height and number of amputations
Patients survival | Three months after drug administration
  Survival

CONTACTS AND LOCATIONS:
Overall Officials: Amir Herman, MD, PhD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Dunser MW, Mayr AJ, Tur A, Pajk W, Barbara F, Knotzer H, Ulmer H, Hasibeder WR. Ischemic skin lesions as a complication of continuous vasopressin infusion in catecholamine-resistant vasodilatory shock: incidence and risk factors. Crit Care Med. 2003 May;31(5):1394-8. doi: 10.1097/01.CCM.0000059722.94182.79. PMID 12771608
- [Background] Fregene A, Ditmars D, Siddiqui A. Botulinum toxin type A: a treatment option for digital ischemia in patients with Raynaud's phenomenon. J Hand Surg Am. 2009 Mar;34(3):446-52. doi: 10.1016/j.jhsa.2008.11.026. PMID 19258141
- [Background] Golbranson FL, Lurie L, Vance RM, Vandell RF. Multiple extremity amputations in hypotensive patients treated with dopamine. JAMA. 1980 Mar 21;243(11):1145-6. PMID 7359665
- [Background] Van Beek AL, Lim PK, Gear AJL, Pritzker MR. Management of vasospastic disorders with botulinum toxin A. Plast Reconstr Surg. 2007 Jan;119(1):217-226. doi: 10.1097/01.prs.0000244860.00674.57. PMID 17255677
- [Background] Janz BA, Thomas PR, Fanua SP, Dunn RE, Wilgis EF, Means KR Jr. Prevention of anastomotic thrombosis by botulinum toxin B after acute injury in a rat model. J Hand Surg Am. 2011 Oct;36(10):1585-91. doi: 10.1016/j.jhsa.2011.07.008. Epub 2011 Aug 19. PMID 21855233
- [Background] Clemens MW, Higgins JP, Wilgis EFS. Prevention of anastomotic thrombosis by botulinum toxin a in an animal model. Plast Reconstr Surg. 2009 Jan;123(1):64-70. doi: 10.1097/PRS.0b013e3181904c31. PMID 19116537